CLINICAL TRIAL: NCT04345835
Title: Prone Flexed Position in Percutanous Nephrolithotomy in Comparsion With Standard Prone Position. A Randomized Controlled Trial.
Brief Title: Prone Flexed Position in Percutanous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Diaa Eldin Taha Ramadan Mohamed, Lecturer of urology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS/19.20
Record Dates: First submitted 2020-04-12; First posted 2020-04-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Renal Stones
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prone flexed (Active Comparator): prone flexed PCNL position
  Interventions: Procedure: Percutanous nephrolithotomy (PCNL)
- prone (Active Comparator): prone position PCNL
  Interventions: Procedure: Percutanous nephrolithotomy (PCNL)

INTERVENTIONS:
Procedure: Percutanous nephrolithotomy (PCNL) — different procedure positioning
  Other Names: PNL

SUMMARY:
prone flexed position in percutanous nephrolithotomy in comparsion with standard prone position. A randomized controlled trial.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will be randomly allocated to 2 groups:

1. 1st group will undergo prone-flexed PCNL.
2. 2nd group will undergo prone PCNL.

III. Recruitment of participants Patients appointed for an outpatient diagnostic cystoscopy will be reviewed for the inclusion and exclusion criteria. Legible patients will be asked to participate in the study and to sign the informed consent form.

IV. Randomisation Randomization will be performed using computer generated random tables using stratified blocked randomization in 1:1 ratio.

V. Study procedure Preoperative evaluations included

1. Detailed medical history
2. Physical examination
3. Routine blood examination
4. Urinalysis & urine cytology
5. Renal and liver function tests
6. Coagulation profile

8. Computed tomography of the abdomen and pelvis

Operative Technique

Prone-flexed positioning i. Retrograde access will be obtained ii. The patient is repositioned prone with adequate padding under the pressure points of the head, chest, knees, and feet.

iii. The table is flexed 30 degrees at the level of the patient's mid lumbar region to open the space between the 12th rib and the posterior iliac crest dropping the gluteal muscles from the working plane.

Ancillary intervention

Patients will receive a 20-mL infiltration of 0.25% bupivacaine. Under fluoroscopic guidance, the local analgesic was infiltrated with a 22-gauge spinal needle (10-cm length) along the nephrostomy tract at the 3, 6, 9, and 12 o'clock positions (5 mL in each tract), including the muscles, subcutaneous tissue, and skin.

Patients will receive 1 g tranexamic acid at induction followed by three further doses of 500 mg over the next 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Large renal or upper ureteral calculi or both,

Exclusion Criteria:

* (1) Age <18 years or Pregnancy (2) Ureter pelvic junction obstruction (3) Bilateral simultaneous PCNL (4) Need for 3 percutaneous tracts intraoperative (5) Morbid obesity (BMI >40) (6) Non opaque renal stones. (7)Refuse to complete study requirements (8)Untreated UTI (9)Atypical bowel interposition by CT (10)Tumour in the presumptive access tract area or Potential malignant kidney tumour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
position complications | end of the study
  Comparing the prone with the prone-flexed position for PCNL reporting complications using the Clavien-Dindo system

SECONDARY OUTCOMES:
stone score system | end of the study
  Comparison of the Guy's (19)" combines the number of stones, their location, and abnormal patient anatomy into a score 1-4", S.T.O.N.E. (20)"uses the stone size, tract length, obstruction, number of calyces involved, and stone density from patient's preoperative CT scan", and CROES (21) "a continuous variable calculated by stone characteristics, patient data, and surgeon/centre experience" Scores for predicting outcomes following PCNL
stone characteristics | end of the study
  Explore the relationship between stone density using various HU values "highest HU value (HUmax), lowest HU value (HUmin) and average HU value (HUave)"on and outcomes of percutaneous nephrolithotomy (PCNL)
stone volume | end of the study
  Assess the impact of the ellipsoid volume of the stone [volume = π/6*(AP*H*CC)] after measuring the antero-posterior and horizontal dimensions in the axial images and the cranio-caudal dimension in the coronal images on and outcomes of percutaneous nephrolithotomy (PCNL).
hemostatic measures | end of the study
  Investigate the effect of antifibrinolytic tranexamic acid usage on blood loss during PCNL.

CONTACTS AND LOCATIONS:
Overall Officials: Diaa Eldin Taha, MD, Principal Investigator — Lecturer of urology
Locations (1):
- Kafrelsheikh faculty of medicine, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No